CLINICAL TRIAL: NCT05372341
Title: Postoperative Outcomes of Covid-19 Patients Who Were Hospitalized in a Training and Research Hospital, Who Were Operated on Electively
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Senay Canikli, Consultant of Anesthesiology, Samsun University
Other Study IDs: GOKA/2021/14/7
Record Dates: First submitted 2022-05-10; First posted 2022-05-12 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Long-term Consequences of COVID-19 Infection
Keywords: Covid-19; postoperative care; elective surgergy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post-covid elective surgery patients: data of postcovid patients underwent elective surgery will be collected.
  Interventions: Other: descriptive

INTERVENTIONS:
Other: descriptive — posotcovid patients will be elective surgery postoperative outcomes

SUMMARY:
The Covid-19 infection has led to global health crisis. As the number of patients recovering from Covid-19 infection increases, it is necessary to create an understanding of the health problems that concern them. Reports of persistent and long-lasting effects are increasing after Covid-19 infection .

DETAILED DESCRIPTION:
Data on postoperative outcomes in the patient population with Covid-19 infection are limited. In more than half of these patients, pulmonary complications and mortality are seen between 19-24%. Covid-19 infection positivity has been shown as an independent risk factor for surgical mortality. In this study, we aimed to examine the results of patients who were hospitalized and operated electively after they has Covid-19. Among the patients who were hospitalized and followed up in our hospital due to Covid-19 infection between July 2020 and July 2021, those over the age 18 and opereted on electively will be included in the study. By accessing the hospital records, patients Covid-19 treatment records, length of hospital stay, intensive care follow-up, processes, pulmonary support conditions, lung involvement, time until the operation, operation type, operation time, ASA classification, anesthesia type, post-operative follow-up processes, post-operation intensive care needs, time to discharge and mortality will be examined. After the data of of the patients were recorded using SPSS19 program, statistical analysis will be performed using the arithmetic mean, median, standart deviation and Chi-square test, which are among the measures of distribution and prevalence.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* those who elective surgery
* patients who have had Covid-19

Exclusion Criteria:

* emergency surgery
* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the files of the patients who were hospitalized in the hospital and who had an additional operation, among the patients who had Covid-19, will be reviewed retrospectively
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
need for postoperative intensive care | 8 months
  after covid-19, the need for postoperative intensive care unit is higer, especially due to pulmonary complications.
prolongation of postoperative hospital stay | 8 months
  longer hospital stay, especially due to pulmonary complications

SECONDARY OUTCOMES:
anesthesia preference status; general or spinal | 8 months
  more regional anesthesia techniques are preferred due to increased risk of pulmonary complications after Covid-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Canikli Adıgüzel, Study Director — responsibl investigator; şenay canikli adıgüzel, Principal Investigator — project manager
Locations (1):
- SAMSUN UNIVERSITY Samsun Training and research hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
personal data of participants will not be shared. Patient files will be coded by giving sequence numbers